CLINICAL TRIAL: NCT02854059
Title: A Phase II Pilot Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacodynamics and Pharmacokinetics of IdeS in Asymptomatic Antibody-Mediated Thrombotic Thrombocytopenic Purpura (TTP) Patients With Low ADAMTS13 Activity
Brief Title: IdeS in Asymptomatic Antibody-Mediated Thrombotic Thrombocytopenic Purpura (TTP) Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor review of initial results demonstrates a non-favourable risk benefit
Sponsor: Hansa Biopharma AB (Industry)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15-HMedIdeS-08
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Purpura, Thrombotic Thrombocytopenic
Keywords: Asymptomatic antibody-mediated TTP
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment IdeS (0.25 mg/kg) (Experimental): A single 30 minutes i.v. infusion of IdeS (0.25 mg/kg). Following an evaluation of safety and efficacy in 3 patients receiving 0.25 mg/kg there will be a potential to increase the IdeS dose to 0.5 mg/kg for the remaining 3 patients.
  Interventions: Biological: IdeS (0.25 mg/kg)
- Treatment IdeS (0.50 mg/kg) (Experimental): A single 30 minutes i.v. infusion of IdeS (0.50 mg/kg).
  Interventions: Biological: IdeS (0.50 mg/kg)

INTERVENTIONS:
Biological: IdeS (0.25 mg/kg) — Single i.v. infusion of IdeS (0.25 mg/kg). Following an evaluation of efficacy and safety in the first 3 patients the dose may be increased in the following 3 patients to 0.5 mg/kg.
  Other Names: HMed-IdeS, IgG-degrading enzyme of Streptococcus pyogenes
  Arms: Treatment IdeS (0.25 mg/kg)
Biological: IdeS (0.50 mg/kg) — Single i.v. infusion of IdeS (0.50 mg/kg).
  Other Names: HMed-IdeS, IgG-degrading enzyme of Streptococcus pyogenes
  Arms: Treatment IdeS (0.50 mg/kg)

SUMMARY:
The main purpose of this study is to evaluate safety and tolerability in patients diagnosed with asymptomatic antibody-mediated TTP with low ADAMTS13 activity after receiving single intravenous dose of IdeS.

DETAILED DESCRIPTION:
Immunoglobulin G-degrading enzyme of Streptococcus pyogenes (IdeS) is an IgG specific endopeptidase which cleaves IgG molecules and efficiently neutralizes Fc-mediated activities. IdeS-mediated IgG degradation constitutes a novel therapeutic principle for the treatment of IgG-driven human diseases.

In addition to assessing the safety and tolerability of IdeS the study will also assess the efficacy of IdeS to significantly increase the ADAMTS13 activity and decrease the anti-ADAMTS13 antibody levels in patients diagnosed with asymptomatic antibody-mediated TTP with low ADAMTS13 activity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Diagnosed with acquired TTP with ADAMTS13 levels of ≤ 10 % in clinical remission and with measurable or previously confirmed ADAMTS13 antibodies

Exclusion Criteria:

* Prior malignancy within 5 years
* Test positive for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus (HIV)
* Ongoing infectious disease including P-CRP >10
* Test positive for IgE antibodies against IdeS
* Secondary cause of TTP
* Rituximab treatment or other antibody-based therapy within 7 days prior to IdeS dosing
* Treatment with investigational medicinal product within the last 12 weeks proceeding screening
* Severe other conditions requiring treatment and close monitoring, e.g. cardiac failure > NYHA (New York Heart Association) grade 3, unstable coronary disease or oxygen dependent COPD
* History of any other clinically significant disease or disorder which may either put the patient at increased risk because of participation in the study, or influence the results or the patient's ability to participate in the study
* Hypogammaglobulinemia defined as any values of P-total IgG less than 3 g/L
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to IdeS (e. g. streptokinase and/or staphylokinase)
* Substance abuse or other concurrent medical condition that could confound study interpretation or affect the patient's ability to tolerate or complete the study
* Breast feeding women or women with a positive pregnancy test
* Previously received IdeS treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Sonesson, PhD, Study Director — Hansa Biopharma AB
Locations (1):
- University College London Hospitals NHS, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
An internal monitoring committee (IMC) at the sponsor will review available safety and tolerability data after 3 patients have received a dose of 0.25 mg/kg before proceeding to the next dose (0.5 mg/kg). Safety data collected up to and including day 14 will be evaluated.

REFERENCES:
- [Derived] Stubbs MJ, Thomas M, Vendramin C, Sonesson E, Kjellman C, Jarnum S, Stenberg Y, Elfving C, Scully M. Administration of immunoglobulin G-degrading enzyme of Streptococcus pyogenes (IdeS) for persistent anti-ADAMTS13 antibodies in patients with thrombotic thrombocytopenic purpura in clinical remission. Br J Haematol. 2019 Jul;186(1):137-140. doi: 10.1111/bjh.15706. Epub 2018 Nov 29. No abstract available. PMID 30488420

RESULTS

PARTICIPANT FLOW:
Groups:
- IdeS (0.50 mg/kg): A single 30 minutes i.v. infusion of IdeS (0.50 mg/kg).
Period: Overall Study
Arm/Group | Treatment IdeS (0.25 mg/kg) | IdeS (0.50 mg/kg)
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: After review of the initial results from the study that demonstrated a non-favourable risk-benefit profile in the first 2 patients who received single i.v. infusion of IdeS (0.25 mg/kg), the study was prematurely discontinued. The potential dose escalation to i.v. infusion of IdeS (0.5 mg/kg) did not occur.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment IdeS (0.25 mg/kg) | Treatment IdeS (0.50 mg/kg) | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Measured by Type, Frequency and Intensity of Adverse Events
Description: Data on AEs were obtained if spontaneously reported by the patient, if reported in response to an open question from the study personnel or if revealed by observation.
  A treatment emergent AE (TEAE) is defined as any AE occurring after administration of the IMP and within the time of the residual drug effect period (i.e. 30 days after IMP administration).
  AEs reported in ClinicalTrials.gov include TEAEs and post-treatment AEs, i.e. all AEs occurring after administration of IdeS until end of study.
  Please refer to Adverse Event section for details on reported AEs
Time Frame: From dosing until end of follow up on day 64
Population: Because of the premature termination of the study due to the non-favourable risk-benefit profile in the first 2 patients and since the sponsor will no longer pursue the indication, the analyses as described in the protocol were not performed. Instead, data collected for the 2 enrolled subjects were listed and/or presented graphically.
Measure: Number; unit: Adverse Events
Arm/Group | Treatment IdeS (0.25 mg/kg) | Treatment IdeS (0.50 mg/kg)
Number analyzed (Participants) | 2 | 0
Adverse Events
  TEAEs | 10 |
  Mild TEAEs (Grade=1) | 7 |
  Moderate TEAEs (Grade=2) | 1 |
  Severe TEAEs (Grade=3) | 1 |
  Life threatening TEAEs (Grade=4) | 1 |
  Related TEAEs | 4 |
  Serious TEAEs | 2 |
  Post-TEAEs | 2 |
  Mild Post-TEAEs (Grade=1) | 1 |
  Moderate Post-TEAEs (Grade=2) | 1 |
  Related Post-TEAEs | 0 |
  Serious Post-TEAEs | 2 |

2. Secondary Outcome: Number of Patients With Change From Baseline in ADAMTS13 Activity
Description: ADAMTS13 is an enzyme which is inhibited in patients with TTP. The efficacy of IdeS on ADAMTS13 activity was measured througout the study as change from baseline.
Time Frame: From day of dosing until end of follow up on day 64
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment IdeS (0.25 mg/kg) | Treatment IdeS (0.50 mg/kg)
Number analyzed (Participants) | 2 | 0
Participants
  Change in ADAMTS13 at any timepoint after IdeS | 0 |
  No change in ADAMTS13 at any time after IdeS | 2 |

3. Secondary Outcome: Number of Patients With Change From Baseline in ADAMTS13 Antibody Levels
Description: The efficacy of IdeS on ADAMTS13 antibody cleaving was measured througout the study as change from baseline in ADAMTS13 antibody concentration.
Time Frame: From day of dosing until end of follow up on day 64
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment IdeS (0.25 mg/kg) | Treatment IdeS (0.50 mg/kg)
Number analyzed (Participants) | 2 | 0
Participants
  ≥90% decrease in antibodies 2-24h after IdeS | 2 |
  <90% decrease in antibodies 2-24h after IdeS | 0 |

4. Secondary Outcome: Number of Patients for Whom a Decreased ADAMTS13 Activity Returned to Normal Levels at Different Time-points in the Study
Description: The ADAMTS13 activity in TTP patients is decreased. The efficacy of IdeS on ADAMTS13 activity was assessed throughout the study to identify the time-point of return to normal levels.
Time Frame: From day of dosing until end of follow up on day 64
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment IdeS (0.25 mg/kg) | Treatment IdeS (0.50 mg/kg)
Number analyzed (Participants) | 2 | 0
Participants
  Normal ADAMTS13 activity any time after IdeS | 0 |
  Decreased ADAMTS13 activity all time after IdeS | 2 |

5. Secondary Outcome: Number of Patients With Change From Baseline in Pharmacodynamics as Measured by Level of IgG
Description: IdeS cleaves IgG molecules. The concentration of uncleaved IgG in the patient's serum was measured throughout the study to determine change from baseline following IdeS administration.
Time Frame: From day of dosing until end of follow up on day 64
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment IdeS (0.25 mg/kg) | Treatment IdeS (0.50 mg/kg)
Number analyzed (Participants) | 2 | 0
Participants
  ≥90% decrease in IgG 2-24h after IdeS | 2 |
  ≥90% decrease in IgG 3 days after IdeS | 1 |
  ≥90% decrease in IgG 7-64 days after IdeS | 0 |

6. Secondary Outcome: Number of Patients Showing IdeS Immunogenicity as Measured by Anti-drug Antibodies
Description: Most humans have been infected with S. pyogenes which is the origin of IdeS. It was therefore expected that patients in this study might have antibodies against IdeS before being exposed to IdeS in the study. The concentration of ant-IdeS antibodies was measured before dosing and throughout the study.
Time Frame: From day of dosing until end of follow up on day 64
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment IdeS (0.25 mg/kg) | Treatment IdeS (0.50 mg/kg)
Number analyzed (Participants) | 2 | 0
Participants
  Presence of anti-IdeS antibodies before IdeS | 2 |
  Elevated anti-IdeS antibodies Day 64 | 2 |

7. Secondary Outcome: Maximum Serum Concentration (Cmax) of IdeS
Description: The concentration of IdeS in serum was measured to identify the pharmacokinetic parameter Cmax of IdeS in TTP patients.
Time Frame: From day of dosing until day 14
Population: Because of the premature termination of the study due to the non-favourable risk-benefit profile in the first 2 patients and since the sponsor will no longer pursue the indication, the analyses as described in the protocol were not performed. Instead, data collected for the 2 enrolled subjects were listed and presented graphically.
Measure: Mean (Full Range); unit: µg/mL
Arm/Group | Treatment IdeS (0.25 mg/kg) | Treatment IdeS (0.50 mg/kg)
Number analyzed (Participants) | 2 | 0
µg/mL | 6.64 [4.60 to 8.67] |

8. Secondary Outcome: Time-point for Maximum Serum Concentration of IdeS
Description: The concentration of IdeS in serum was measured to identify the pharmacokinetic parameter Tmax of IdeS in TTP patients. Tmax refers to the time-point when the serum concentration of IdeS reaches maximum.
Time Frame: From day of dosing until day 14
Population: as for outcome 7
Measure: Mean (Full Range); unit: hours
Arm/Group | Treatment IdeS (0.25 mg/kg) | Treatment IdeS (0.50 mg/kg)
Number analyzed (Participants) | 2 | 0
hours | 1.38 [0.75 to 2.00] |

9. Secondary Outcome: Number of Patients With Change From Baseline in Pharmacodynamics as Measured by Level of F(ab')2 Fragments
Description: The efficacy of IdeS can be measured as change from baseline in F(ab')2 fragments (i.e. the antigen binding fragment of IgG).
Time Frame: From day of dosing until end of follow up on day 64
Population: The concentration of F(ab')2 fragments in the patients' serum samples was not analysed because of the premature termination of the study due to the non-favourable risk-benefit profile in the first 2 patients and since the sponsor will no longer pursue the indication.
Arm/Group | Treatment IdeS (0.25 mg/kg) | Treatment IdeS (0.50 mg/kg)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for a time-period of 3 months for the individual subject (i.e. from the subject signed the informed consent form (ICF) throughout the study including the follow-up period until the end of study visit).
Description: Data on AEs were obtained if spontaneously reported by the patient, if reported in response to an open question from the study personnel or if revealed by observation.
  A treatment emergent AE (TEAE) was defined as any AE occurring after administration of IdeS and within the time of the residual drug effect period (i.e. 30 days after IdeS administration).
  AEs reported in ClinicalTrials.gov include TEAEs and post-TEAEs, i.e. all AEs occurring after administration of IdeS until end of study
Arm/Group | Treatment IdeS (0.25 mg/kg) | Treatment IdeS (0.50 mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment IdeS (0.25 mg/kg) (N=2) | Treatment IdeS (0.50 mg/kg) (N=0)
Serum sickness (Immune system disorders) | 2 (2) | NA
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment IdeS (0.25 mg/kg) (N=2) | Treatment IdeS (0.50 mg/kg) (N=0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | NA
Pyrexia (General disorders) | 1 (2) | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | NA
Headache (Nervous system disorders) | 1 (1) | NA
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | NA
Tachycardia (Cardiac disorders) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All MS must be sent to Sponsor for review at least 60d before submission. Sponsor may request changes. All reasonable comments will be incorporated by Investigator. If MS contains info that could impact proprietary or IP interests, the Sponsor is entitled to request a 6 mth publication delay, allowing actions to protect its interests. The Investigator/Trust shall not unreasonably withhold or delay its consent to such request from the Sponsor or for an exceptional additional delay if requested.

DOCUMENTS (2):
  • Study Protocol (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT02854059/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT02854059/SAP_001.pdf